CLINICAL TRIAL: NCT05515133
Title: Correlation of Psychological Stress With Quality of Life and Efficacy of Immunotherapy Response in Patients With Newly Diagnosed Glioblastoma
Brief Title: Correlation Between Psychological Stress and Disease Progression in Newly Diagnosed Glioblastoma Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HenanPPH-Glioma
Record Dates: First submitted 2022-08-21; First posted 2022-08-25 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-08

CONDITIONS: Glioblastoma
Keywords: glioblastoma; psychological stress; Immune microenvironment
MeSH Terms: conditions — Glioblastoma; Stress, Psychological | interventions — Anthropogenic Effects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observation group of newly diagnosed glioblastoma patients with high-level psychological stress: The patients had high threshold levels of perceived stress, psychological distress, fear, anxiety, and depression as assessed by psychologists
  Interventions: Other: stressors
- Observation group of newly diagnosed glioblastoma patients with low-level psychological stress: The patients had lower than threshold levels of perceived stress, psychological distress, fear, anxiety, and depression as assessed by psychologists

INTERVENTIONS:
Other: stressors — Patients are exposed to stressful situations related to the diagnosis and treatment of the disease
  Groups: Observation group of newly diagnosed glioblastoma patients with high-level psychological stress

SUMMARY:
It is a single-center, prospective, observational，non-randomized study of newly diagnosed glioblastoma patients conducted in a tertiary hospital. The investigators examine the psychological stress, immune biomarker changes, quality of life, and disease progression of patients with glioblastoma at five-time points.

The study had two cohorts, a high-stress cohort and a low-stress cohort, which are grouped after initial recruitment. Both groups undergo total resection of tumors and received 3 months of standardized treatment with radiotherapy and chemotherapy. Neither participants nor doctors but the researcher can choose which group participants are in. No one knows if one study group is better or worse than the other.

DETAILED DESCRIPTION:
Glioblastoma (GBM) is the most common and aggressive primary malignant brain tumor affecting adults, with a median survival of 12-16 months after diagnosis. The diagnosis of a malignant tumor has a huge impact on patients' psychology, which is easy to lead to patients in a state of stress.

The high-stress level can lead to a change in patients' health behaviors and correlates with the prognosis outcome. In addition, psychological stress can lead to changes in the immune microenvironment, but disease progression and quality of life in glioblastoma have not been adequately demonstrated.

Grouping process: 60 patients are expected to be enrolled. After enrollment, participants will receive regular tumor in situ fluid (fluid within the surgical cavity, TISF) sampling for tumor mutation burden（TMB) analysis and recceive regular MRI. Under the standard of care, participants will receive psychological stress assessment after being diagnosed. according to five psychological scales, and the patients were grouped according to the cut-off value of each scale, the psychological stress of the patients is measured by distress thermometer (DT), perceived stress scale (PSS), anxiety/depression (HADS), VAS stress, and fear of disease progression scale（PoP-Q-SF).

Primary study objectives:

• To evaluate the changes in immune markers of acute and chronic psychological stress in patients with glioblastoma after diagnosis.

Secondary study objectives:

* To evaluate the quality of life of patients with different psychological stress levels.
* To evaluate the progression-free survival of patients with different psychological stress levels.

Exploratory objectives:

* To evaluate the effect of managing the patient's psychological stress on the patient's immune microenvironment.
* To evaluate the incidence of mental illness.
* To evaluate the patient treatment compliance.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years
* Karnofsky Performance Score ≥ 70 %
* histologically confirmed, previously untreated GBM
* receiving a standardized chemoradiotherapy regimen
* no previous history of mental illness, drug abuse, or alcohol abuse
* ability to communicate and read and write independently
* willing and able to comply with the protocol as judged by the investigator's signed informed consent.

Exclusion Criteria:

* Patients who have any other disease, either metabolic or psychological, or who have any evidence on clinical examination or special investigations (including laboratory findings) which give reasonable suspicion of a condition that interferes with the adequate measurement of the stress axis (e.g. chronic use of corticosteroids ≥ 3 months before study entry for diseases other than glioblastoma, (dexamethasone use in the context of glioblastoma is allowed) Severe, medically treated psychiatric disorder prior to the diagnosis of glioblastoma Participation in a study with investigational drugs.
* pregnancy or breast-feeding
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, neurologic deficits that interfere with the planned walking tests, dementia, or confusional state.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: newly diagnosed glioblastoma
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-12-15 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor mutation burden（TMB） | From the time of diagnosis to 12 months
  The proportion of tumor mutational burden ≥10 Mut/MB in the population who remain progression-free after diagnosis.
The proportion of patients with high-level psychological stress | From the time of diagnosis to 12 months
  The self-report questionnaire of Perceived Stress Scale（PSS）is used to measure the psychological stress level of patients, with 43 as the critical value, more than or equal to 43 as the high level of psychological stress, less than 43 as the low level of psychological stress.

SECONDARY OUTCOMES:
The Short Form-36 (SF-36) | From the time of diagnosis to 12 months
  The questionnaire of Short Form-36 (SF-36) is used health-related quality-of-life measure in participants outcomes. The scale contains 9 dimensions with a total score of 100 points.
Progression-free survival at 6 months | From the time of diagnosis to 12 months
  The proportion of participants in the analysis population who remain progression-free for at least six months after diagnosis.

OTHER OUTCOMES:
Overall survival rate at 12 months | From the time of diagnosis to 12 months
  OS-12 is the proportion of participants in the analysis population who remain alive for at least twelve months after diagnosis.
Progression-free survival | Up to 3 years after diagnosis
  Median time from allocation to first documented disease progression as per RANO or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Xingyao Bu, MD, Study Director — Henan Provincial People's Hospital; Jie Mei, MD, Principal Investigator — Henan Provincial People's Hospital
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No